CLINICAL TRIAL: NCT04239365
Title: Follow-up Protocol of Colorectal Endoscopic Mucosal Resection Scars: a Multicentre Randomized Single-blinded Crossover Trial
Brief Title: Follow-up Protocol of Colorectal Endoscopic Mucosal Resection Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portuguese Oncology Institute, Coimbra (Other)
Responsible Party: Principal Investigator, Mafalda Cainé João, Medical Doctor, Portuguese Oncology Institute, Coimbra
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PortugueseOIC 004
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer; Recurrence, Local Neoplasm
Keywords: recurrence; endoscopic mucosal resection; colorectal lesions; advanced endoscopic imaging
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Recurrence, Local; Recurrence

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: WLE followed by NBI (Experimental): EMR scar is interrogated using WLE followed by NBI
  Interventions: Diagnostic Test: WLE followed by NBI or NBI followed by WLE (crossover design)
- Group B: NBI followed by WLE (Active Comparator): EMR scar is interrogated using NBI followed by WLE
  Interventions: Diagnostic Test: WLE followed by NBI or NBI followed by WLE (crossover design)

INTERVENTIONS:
Diagnostic Test: WLE followed by NBI or NBI followed by WLE (crossover design) — EMR scar is inspected using WLE followed by NBI or vice versa
  Other Names: WLE followed by NBI or NBI followed by WLE

SUMMARY:
Nowadays endoscopic mucosal resection (EMR) is the gold standard for the removal of large laterally spreading and sessile colorectal lesions ≥ 20 mm. However, recurrence rate after successful EMR (defined by the absence of neoplastic tissue at the completion of the procedure after careful inspection of the post-EMR mucosal defect and margin) is about 15-20%. Consequently, current guidelines recommend a surveillance colonoscopy between 4 and 6 months after resection for detection of residual or recurrent polyp.

There are few studies that have examined the accuracy of advanced endoscopic imaging for the prediction of histological recurrence but none of these imaging modalities have been validated for surveillance after EMR. Therefore, current guidelines strongly recommend systematic biopsy of EMR scar.

The main aim of this study is to assess the incremental benefit of narrow band imaging (NBI) and white light endoscopy (WLE) randomizing the initial technique for the endoscopic detection of post-EMR recurrence and to asses if this advanced imaging method achieve sufficient diagnostic accuracy to exclude recurrence without the need for biopsy.

DETAILED DESCRIPTION:
a. Study type: multicenter randomized crossover trial: i. prospective inclusion of consecutive patients undergoing first follow-up surveillance colonoscopy after successful EMR of colorectal lesion; ii. crossover randomization by computer generated tables; iii. allocation concealment by sealed, opaque envelopes; iv. pathologist-blinded - pathologists are blinded to the study protocol and samples are received as 'EMR scar for assessment' .

b. Selection patient method: inclusion by invitation of patients undergoing the first follow-up surveillance colonoscopy after successful EMR of colorectal lesion.

c. Sample size: 210 (two groups of 105 patients). To improve accuracy from 85% (value obtained by a study that did not show significant differences in the accuracy of NBI followed by WLE vs. WLE followed by NBI) to 95% and assuming a normal distribution and a power of 80% (α=0.05), the calculated sample size of each of the 2 groups was 96; allowing for a 10% dropout rate, the sample size is 105 per group (210 patients overall).

d. Procedures and data collection methods: i. Each procedure is performed by the same endoscopist. ii. All patients receive split dose bowel preparation. iii. All colonoscopies are performed using high definition colonoscopes with NBI ( EVIS EXERA III CV 185 and CV 190; Olympus Inc., Tokyo, Japan). iv. Colon inspection is done with WLE during withdrawal. v. At the proximity of the scar WLE and NBI were used randomly one after the other (WLE>NBI or NBI>WLE). If NBI is the first technique used, it is switched prior to scar detection, avoiding, as far as possible, a glance with WLE. The edges of the scar are interrogated followed by the centre of the scar and finding are recorded. vi. After both evaluations, if there is no suspicion of recurrence, the site is sampled by at least 2 biopsies of the scar edge. If there is any suspicion of recurrence, tissue sample is obtained and then treated by endoscopic resection using standard methods. At least 2 biopsies specimens from normal appearing scar are also obtained.

e. Analysed variables: i. patient characteristics; ii. data from baseline colonoscopy; iii. data from first surveillance colonoscopy (see outcome measures).

f. Statistical analysis: i. Performed using statistical software IBM SPSS Statistics, Version 25.0. Armonk, NY: IBM Corp. ii. Continuous variables are reported as mean and standard deviation or median and interquartile range, if they have normal or not normal distribution, respectively; categorical variables as absolute and relative frequency. iii. Continuous variables are compared between two groups using Student's T test if they have a normal distribution and homogeneity of variance or Mann-Whitney U if these conditions are not met. Categorical variables are compared using Pearson's X2 test or Fisher test. iv. Sensitivity, specificity, negative and positive predictive values and accuracy are calculated using 2x2 contingency tables. v. All hypotheses are two-tailed and a P-value<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing the first follow-up surveillance colonoscopy after successful EMR of colorectal lesion.

Exclusion Criteria:

* informed consent not provided,
* inflammatory bowel disease, inadequate bowel preparation (Boston Bowel Preparation Scale total score < 6 or < 2 in a segment),
* EMR scar not identified during colonoscopy,
* tissue acquisition unfeasibly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of WLE and NBI for each group | 1 day (at the time of data analysis)
  Sensitivity, specificity, negative predictive value, positive predictive value and accuracy of NBI and WLE for each group calculated using 2x2 contingency tables
Recurrent adenoma - WLE | 1 day (during colonoscopy)
  WLE recurrent adenoma identification for each group
Recurrent adenoma - NBI | 1 day (during colonoscopy)
  NBI recurrent adenoma identification for each group
Recurrent adenoma - histology | 1 day (within 30 days from colonoscopy)
  Adenoma recurrence confirmed by histology

SECONDARY OUTCOMES:
Lesion characterization at the baseline colonoscopy | 1 day (at the time of patient inclusion)
  Lesion size and location, Paris classification, NICE classification, number of pieces, use of adjunctive ablative techniques and those identification and histology. Data collected by endoscopic reports consultation
Scar characterization at the first surveillance colonoscopy | 1 day (immediately after first surveillance colonoscopy)
  Scar size, presence or absence of recurrence, in case of recurrence: number of sites, location (edge of the scar, within the scar or both), morphology of recurrence, NICE classification (for NBI evaluation)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Areia, PhD, Study Director — Gastroenterology Department
Locations (1):
- Portuguese Oncology Institute - Coimbra, Coimbra, Portugal

REFERENCES:
- [Background] Rembacken B, Hassan C, Riemann JF, Chilton A, Rutter M, Dumonceau JM, Omar M, Ponchon T. Quality in screening colonoscopy: position statement of the European Society of Gastrointestinal Endoscopy (ESGE). Endoscopy. 2012 Oct;44(10):957-68. doi: 10.1055/s-0032-1325686. Epub 2012 Sep 17. No abstract available. PMID 22987217
- [Background] Tate DJ, Desomer L, Klein A, Brown G, Hourigan LF, Lee EY, Moss A, Ormonde D, Raftopoulos S, Singh R, Williams SJ, Zanati S, Byth K, Bourke MJ. Adenoma recurrence after piecemeal colonic EMR is predictable: the Sydney EMR recurrence tool. Gastrointest Endosc. 2017 Mar;85(3):647-656.e6. doi: 10.1016/j.gie.2016.11.027. Epub 2016 Nov 28. PMID 27908600
- [Background] Hassan C, Quintero E, Dumonceau JM, Regula J, Brandao C, Chaussade S, Dekker E, Dinis-Ribeiro M, Ferlitsch M, Gimeno-Garcia A, Hazewinkel Y, Jover R, Kalager M, Loberg M, Pox C, Rembacken B, Lieberman D; European Society of Gastrointestinal Endoscopy. Post-polypectomy colonoscopy surveillance: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2013 Oct;45(10):842-51. doi: 10.1055/s-0033-1344548. Epub 2013 Sep 12. PMID 24030244
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Desomer L, Tutticci N, Tate DJ, Williams SJ, McLeod D, Bourke MJ. A standardized imaging protocol is accurate in detecting recurrence after EMR. Gastrointest Endosc. 2017 Mar;85(3):518-526. doi: 10.1016/j.gie.2016.06.031. Epub 2016 Jun 22. PMID 27343411
- [Background] Kandel P, Brand EC, Pelt J, Ball CT, Chen WC, Bouras EP, Gomez V, Raimondo M, Woodward TA, Wallace MB; EMR SCAR Group. Endoscopic scar assessment after colorectal endoscopic mucosal resection scars: when is biopsy necessary (EMR Scar Assessment Project for Endoscope (ESCAPE) trial). Gut. 2019 Sep;68(9):1633-1641. doi: 10.1136/gutjnl-2018-316574. Epub 2019 Jan 11. PMID 30635409
- [Background] Riu Pons F, Andreu M, Gimeno Beltran J, Alvarez-Gonzalez MA, Seoane Urgorri A, Dedeu JM, Barranco Priego L, Bessa X. Narrow band imaging and white light endoscopy in the characterization of a polypectomy scar: A single-blind observational study. World J Gastroenterol. 2018 Dec 7;24(45):5179-5188. doi: 10.3748/wjg.v24.i45.5179. PMID 30568394
- [Background] Hayashi N, Tanaka S, Hewett DG, Kaltenbach TR, Sano Y, Ponchon T, Saunders BP, Rex DK, Soetikno RM. Endoscopic prediction of deep submucosal invasive carcinoma: validation of the narrow-band imaging international colorectal endoscopic (NICE) classification. Gastrointest Endosc. 2013 Oct;78(4):625-32. doi: 10.1016/j.gie.2013.04.185. Epub 2013 Jul 30. PMID 23910062
- [Background] The Paris endoscopic classification of superficial neoplastic lesions: esophagus, stomach, and colon: November 30 to December 1, 2002. Gastrointest Endosc. 2003 Dec;58(6 Suppl):S3-43. doi: 10.1016/s0016-5107(03)02159-x. No abstract available. PMID 14652541
- [Derived] Joao M, Areia M, Pinto-Pais T, Gomes LC, Saraiva S, Alves S, Elvas L, Brito D, Saraiva S, Teixeira-Pinto A, Claro I, Dinis-Ribeiro M, Cadime AT. Can white-light endoscopy or narrow-band imaging avoid biopsy of colorectal endoscopic mucosal resection scars? A multicenter randomized single-blind crossover trial. Endoscopy. 2023 Jul;55(7):601-607. doi: 10.1055/a-2018-1612. Epub 2023 Jan 23. PMID 36690030